CLINICAL TRIAL: NCT04929093
Title: Comparative Study of Novel and Conventional Dose Adjustment Schedules for Late Injection of More Than 16 Weeks in Subcutaneous Immunotherapy in Allergic Rhinitis
Brief Title: Novel Dose Adjustment Schedule for Late Injection in SCIT in AR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-SIT-16w
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Allergic Rhinitis; Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Novel dose adjustment schedule (Experimental): The patients in this group had late injections of more than 16 weeks in maintenance period, and restarted SCIT with novel dose adjustment schedule.
  Interventions: Biological: Novel dose adjustment of Alutard SQ
- Conventional dose adjustment (Active Comparator): The patients in this group had late injections of more than 16 weeks in maintenance period, and restarted SCIT with conventional dose adjustment schedule.
  Interventions: Biological: conventional dose adjustment of Alutard SQ
- Continuous cluster SCIT schedule (Active Comparator): The subjects had a routine cluster SCIT schedule without interrupted period.
  Interventions: Biological: Routine continuous cluster of Alutard SQ

INTERVENTIONS:
Biological: Novel dose adjustment of Alutard SQ — novel dose adjustment schedule means directly reaching dose of Vial 4, 10,000 SQ
  Arms: Novel dose adjustment schedule
Biological: conventional dose adjustment of Alutard SQ — conventional dose adjustment schedule means restarting from dose of Vial 1, 10 SQ
  Arms: Conventional dose adjustment
Biological: Routine continuous cluster of Alutard SQ — Patient receiving continuous cluster SCIT for DM during the same period
  Arms: Continuous cluster SCIT schedule

SUMMARY:
Allergen specific immunotherapy is currently the only curative intervention for allergic rhinitis (AR). Subcutaneous immunotherapy (SCIT) need to be reinstituted with an interruption of more than 16 weeks in maintenance period, leading to increased time and economic cost burden and difficulties for continuing further treatment for patients. The aim of present study was to develop a novel dose adjustment schedule for such situation and to compare the clinical efficacy and adverse reactions between novel and conventional schedules for dust mite (DM) SCIT of AR subjects.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18 to 60 years;
* (2) only had a positive response to Der p and Der f but no other inhalant allergens based on EUROline Allergy Diagnostics (Beijing Oumeng Biotechnology Co., Ltd., Beijing, China). Meanwhile at least Der p -specific IgE (sIgE) in serum of was ≥ 0.7 kU/l (CAP Pharmacia, Uppsala, Sweden) using ImmunoCAP system (Pharmacia, Uppsala, Sweden) regardless of the result of Der p -specific IgE in serum;
* (3) had reached cluster SCIT maintenance period and the overall treatment time was more than 1 year but less than 2 years;
* (4) hope to continue to complete the entire treatment and have good compliance.

Exclusion Criteria:

* (1) diagnosed as asthma based on the guidelines of the Global Initiative for Asthma(13);
* (2) had Grade II or above systemic adverse reactions occurred in the past SCIT period.

Ages: 5 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The change of Combined Symptom and Medication Score | baseline, week 3, week 6, week 26.
  CSMS which was calculated as follows: (total nasal symptom scores (TNSS))/4+ MS as recommended by European Academy of Allergy and Clinical Immunology (EAACI) Position Paper. The CSMS score was 0-6, 0 for good therapeutic effect and 6 for poor therapeutic effect.

SECONDARY OUTCOMES:
The change of total nasal symptom scores | baseline, week 3, week 6, week 26.
  last 7 days' overall symptom scores of major nasal symptoms (nasal obstruction, nasal itching, sneezing, and rhinorrhea: 0, no symptoms; 1, mild; 2, moderate; 3, serious). TNSS scores was 0 to 12 (0 = no symptoms;12 = most severe symptoms).
The change of medication score | Baseline, week 26.
  MS was calculated as follows: 1, oral Clarityne tablet; 2, intranasal Budesonide nasal spray.
Adverse reactions | week 26.
  The patients were instructed to immediately report to the physician if any symptom appeared or adverse reactions occurred during the observation period. The time and severity of onset, estimation of a possible reason, resolution, and outcome should be recorded. The adverse reactions were classified in terms of the localization (local or systemic) and the time of appearance (immediate or delayed). Local reactions (LRs) were expressed as the length of the wheal diameter. Systemic reactions (SRs) were graded in accordance with the standards of the EAACI

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tongren Hospital, China
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China